CLINICAL TRIAL: NCT04035226
Title: A Prospective, Multinational Study of Real-life Current Standards of Care in Patients With Relapsed and/or Refractory Multiple Myeloma Who Received at Least 3 Prior Lines of Therapy Including PI, IMID, and CD38 Monoclonal Antibody Treatment
Brief Title: A Study of Real-life Current Standards of Care in Patients With Relapsed and/or Refractory Multiple Myeloma Who Received at Least 3 Prior Lines of Therapy Including Proteasome Inhibitor (PI), Immunomodulatory Drug (IMID), and Cluster of Differentiation 38 (CD38) Monoclonal Antibody Treatment
Acronym: LocoMMotion
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Collaborators: Legend Biotech (Unknown)
Responsible Party: Sponsor
Other Study IDs: CR108651; 68284528MMY4001 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsed/refractory Multiple Myeloma: Patients with relapsed/refractory multiple myeloma who received at least 3 prior lines of therapy including Proteasome Inhibitor (PI), Immunomodulatory Drug (IMID), and Cluster of Differentiation 38 (CD38) Monoclonal Antibody treatment will be observed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered as a part of this study.

SUMMARY:
The purpose of this study is to assess the safety and clinical response including overall response rate (ORR) of real-life standard-of-care (SOC) treatments under routine clinical practice, over a 24-month period, in patients with relapsed/refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of multiple myeloma according to International myeloma working group (IMWG) diagnostic criteria
* Received at least 3 prior lines of therapy or are double refractory to a proteasome inhibitor (PI) and an immunomodulatory agent (IMID) (induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen). Patients will have undergone at least 1 complete cycle of treatment for each regimen (unless progressive disease was the best response)
* Must have documented evidence of progressive disease based on study physician's determination of response by the IMWG response criteria on or after the last regimen. Patients with documented evidence of progressive disease within the previous 6 months and who are refractory or nonresponsive to their most recent line of treatment afterwards are also eligible
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1
* Must not be pregnant or must not plan to become pregnant within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/refractory multiple myeloma (RRMM) receiving antimyeloma treatment as standard of care (SOC) under routine clinical practice will be observed. The main source of data collection will be medical records of each patient.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  ORR is defined as the percentage of patients who achieve a partial response (PR) or better according to the international myeloma working group (IMWG) response criteria.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) Rate | Up to 24 months
  VGPR rate is defined as the percentage of patients who achieve a VGPR or better according to IMWG response criteria.
Complete Response (CR) Rate | Up to 24 months
  CR rate is defined as the percentage of patients who achieve a complete response (CR) or better according to IMWG response criteria.
Stringent Complete Response (sCR) Rate | Up to 24 months
  sCR rate is defined as the percentage of patients who achieve a stringent complete response (sCR) according to IMWG response criteria.
Minimal Residual Disease (MRD) Negative Rate | Up to 24 months
  Minimal residual disease (MRD) negative rate is defined as the percentage of patients with negative MRD status according to IMWG response criteria.
Clinical Benefit Rate (CBR) | Up to 24 months
  CBR is defined as the percentage of patients with clinical benefit. CBR = ORR (sCR + CR + VGPR + PR) + minimal response (MR).
Duration of Response | Up to 24 months
  Duration of response is defined as time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease (according to IMWG criteria).
Time to Response | Up to 24 months
  Time to response is defined as the time between the date of Day 1 of Cycle 1 and the first clinical response evaluation that the patient has met all criteria for PR or better response.
Time to Next Treatment [TTNT] | Up to 24 months
  Time to next treatment is defined as the time from diagnosis to the start of the next-line treatment.
Progression-free Survival (PFS) | Up to 24 months
  PFS is defined as the time from the date of Day 1 of Cycle 1 to the date of first documented disease progression (according to IMWG response criteria) or death due to any cause, whichever occurs first.
Time to Progression on the Next Line of Subsequent Antimyeloma Therapy or Death (PFS2) | Up to 24 months
  PFS2 is defined as the time from the date of Day 1 of Cycle 1 to progression on the next line of subsequent antimyeloma therapy or death, whichever occurs first.
Overall Survival (OS) | Up to 24 months
  Overall survival is the duration from the date of Day 1 of Cycle 1 to the date of the patient's death or study completion, whichever occurs first.
Change from Baseline in Health-related Quality of Life (HRQoL) using European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Scale Score | Baseline up to 24 months
  The EORTC QLQ-C30 version 3 includes 30 items in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single symptom items. The responses are reported using a verbal rating scale. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater health-related quality-of-life (HRQoL), better functioning, and more (worse) symptoms.
Change from Baseline in Health-related Quality of Life (HRQoL) using European Organization for Research and Treatment of Cancer (EORTC) QLQ-MY20 Scale Score | Baseline up to 24 months
  The EORTC QLQ-MY20 was designed to use alongside the EORTC QLQ-C30 to address issues of more relevance to myeloma patients. Four single items from the EORTC QLQ-MY20 will be performed to assess emotional health status (feel restless or agitated, thinking about your illness, worried about dying, worried about health in the future) on scale of 1 (not at all) to 4 (very much).
Change from Baseline in Health-related Quality of Life (HRQoL) using EQ-5D-5L Questionnaire Score | Baseline up to 24 months
  EuroQol Five Dimension (EQ-5D-5L) is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Number of Patients with Adverse Events (AEs) | Up to 24 months
  An AE is any untoward medical occurrence in a patient participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Severity of Adverse Events as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Up to 24 months
  Severity of AEs has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; Grade 5: Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (75):
- United States (12):
  - Oncology Institute of Hope and Innovation, Glendale, California
  - Marin Cancer Center, Greenbrae, California
  - Asclepes Research, Weeki Wachee, Florida
  - Oncology Hematology Assoc of Central Illinois, P.C. d.b.a. Illinois CancerCare, P.C., Peoria, Illinois
  - Providence Cancer Center, Southfield, Michigan
  - Central Care Cancer Center, Bolivar, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Optum Care, Las Vegas, Nevada
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - The Cancer Institute at St. Francis Hospital, East Hills, New York
  - North Shore Hematology Oncology Associates, P.C., East Setauket, New York
  - The Ohio State University, Columbus, Ohio
- Belgium (4):
  - Grand Hopital de Charleroi, site Notre Dame, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Ucl de Mont-Godinne, Yvoir
- France (9):
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier Régional Universitaire de Lille, Hôpital Claude Huriez, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - C.H.U. Hotel Dieu - France, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Pôle IUC Oncopole CHU, Toulouse
- Germany (6):
  - Universitaetsklinikum Koelnt, Cologne
  - Universitätsklinik Hamburg-Eppendorf - Orthopädische Universitätsklinik und Poliklinik, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Medizinische Klinik A, Münster
  - Klinikum der Eberhard Karls Universitaet Abt fur innere Med II Haematologie Onkologie Germany, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (16):
  - U.O. Ematologia con Trapianto- AOU Policlinico di Bari, Bari
  - U.O. Ematologia Istituto Tumori Giovanni Paolo II, Bari
  - Istituto di Ematologia Seràgnoli azienda ospedaliera univeristaria Policlinico S.Orsola-Malpighi, Bologna
  - Policlinico di Catania, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Azienda Ospedaliera San Martino - IST, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Universita degli Studi di Padova Azienda Ospedaliera di Pa, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Irccs Crob, Rionero in Vulture
  - Università di Roma La Sapienza, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Cardinale G. Panico, Tricase
  - A.O.U. Citta della Salute e della Scienza di Torino - Presidio Molinette, Turin
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - UMCG, Groningen
  - Erasmus MC - Satellite, Rotterdam
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Szpital Kliniczny im H Swiecickiego Uniwersytetu Medycznego im K Marcinkowskiego w Poznaniu, Poznan
- Russia (3):
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Samara Region Clinical Hospital, Samara
- Spain (13):
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. de Leon, León
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Son Espases, Palma
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Univ. Dr. Peset, Valencia
  - Hosp. Clinico Univ. de Valladolid, Valladolid
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Maidstone Hospital, Kent
  - Kings College Hospital, London
  - St George's Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Marsden NHS Trust Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez Lopez J, Rodriguez-Otero P, Dytfeld D, Jakubowiak A, Schinke C, Besemer B, Anguille S, Manier S, Rasche L, Teipel R, Scheid C, Pawlyn C, Cavo M, Diels J, Ghilotti F, Lau BW, Renaud T, Orel O, Ong F, Ramos DF, Ammann E, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Real-World Physician's Choice of Treatment in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma: Updated Analyses of MonumenTAL-1 vs. LocoMMotion/MoMMent. Adv Ther. 2025 Nov 28. doi: 10.1007/s12325-025-03409-y. Online ahead of print. PMID 41313549
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez-Lopez J, Rodriguez-Otero P, Dytfeld D, Diels J, Strulev V, Haddad I, Renaud T, Ammann E, Cabrieto J, Perualila N, Gan R, Zhang Y, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Current Treatments in the LocoMMotion and MoMMent Studies in Patients with Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Apr;41(4):1576-1593. doi: 10.1007/s12325-024-02797-x. Epub 2024 Feb 24. PMID 38402374
- [Derived] Mateos MV, Weisel K, Diels J, Arribas A, Tamayo M, Schecter JM, Roccia T, Haddad I, Pacaud L, Moreau P. Characterization and Outcomes of Spanish Patients With Relapsed/Refractory Multiple Myeloma Included in the LocoMMotion Study. Clin Lymphoma Myeloma Leuk. 2024 Apr;24(4):224-231.e2. doi: 10.1016/j.clml.2023.12.001. Epub 2023 Dec 7. PMID 38212206
- [Derived] Moreau P, Mateos MV, Gonzalez Garcia ME, Einsele H, De Stefano V, Karlin L, Lindsey-Hill J, Besemer B, Vincent L, Kirkpatrick S, Delforge M, Perrot A, van de Donk NWCJ, Pawlyn C, Manier S, Leleu X, Martinez-Lopez J, Ghilotti F, Diels J, Morano R, Albrecht C, Strulev V, Haddad I, Pei L, Kobos R, Smit J, Slavcev M, Marshall A, Weisel K. Comparative Effectiveness of Teclistamab Versus Real-World Physician's Choice of Therapy in LocoMMotion and MoMMent in Triple-Class Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Feb;41(2):696-715. doi: 10.1007/s12325-023-02738-0. Epub 2023 Dec 19. PMID 38110653
- [Derived] Moreau P, van de Donk NWCJ, Delforge M, Einsele H, De Stefano V, Perrot A, Besemer B, Pawlyn C, Karlin L, Manier S, Leleu X, Weisel K, Ghilotti F, Diels J, Elsada A, Morano R, Strulev V, Pei L, Kobos R, Smit J, Slavcev M, Mateos MV. Comparative Efficacy of Teclistamab Versus Current Treatments in Real-World Clinical Practice in the Prospective LocoMMotion Study in Patients with Triple-Class-Exposed Relapsed and/or Refractory Multiple Myeloma. Adv Ther. 2023 May;40(5):2412-2425. doi: 10.1007/s12325-023-02480-7. Epub 2023 Mar 24. PMID 36961654
- [Derived] Mateos MV, Weisel K, Martin T, Berdeja JG, Jakubowiak A, Stewart AK, Jagannath S, Lin Y, Diels J, Ghilotti F, Thilakarathne P, Perualila NJ, Cabrieto J, Haefliger B, Erler-Yates N, Hague C, Jackson CC, Schecter JM, Strulev V, Nesheiwat T, Pacaud L, Einsele H, Moreau P. Adjusted comparison of outcomes between patients from CARTITUDE-1 versus multiple myeloma patients with prior exposure to proteasome inhibitors, immunomodulatory drugs and anti-CD38 antibody from the prospective, multinational LocoMMotion study of real-world clinical practice. Haematologica. 2023 Aug 1;108(8):2192-2204. doi: 10.3324/haematol.2022.280482. PMID 36546453
- [Derived] Mateos MV, Weisel K, De Stefano V, Goldschmidt H, Delforge M, Mohty M, Cavo M, Vij R, Lindsey-Hill J, Dytfeld D, Angelucci E, Perrot A, Benjamin R, van de Donk NWCJ, Ocio EM, Scheid C, Gay F, Roeloffzen W, Rodriguez-Otero P, Broijl A, Potamianou A, Sakabedoyan C, Semerjian M, Keim S, Strulev V, Schecter JM, Vogel M, Wapenaar R, Nesheiwat T, San-Miguel J, Sonneveld P, Einsele H, Moreau P. LocoMMotion: a prospective, non-interventional, multinational study of real-life current standards of care in patients with relapsed and/or refractory multiple myeloma. Leukemia. 2022 May;36(5):1371-1376. doi: 10.1038/s41375-022-01531-2. Epub 2022 Mar 24. PMID 35332278